CLINICAL TRIAL: NCT05350605
Title: The Effect of Different Breastfeeding Position Education With Lactation Simulation Model on Breastfeeding
Brief Title: The Effect of Breastfeeding Position Education on Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 125
Record Dates: First submitted 2022-03-22; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Breastfeeding Education
Keywords: Breastfeeding Education; Lactation Simulation Model; Nipple problems; Breastfeeding self-efficacy; Breastfeeding success

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Experimental Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Laid back breastfeding position education group (Experimental): Breastfeeding education will be given to pregnant women in the laid-back breastfeeding position group, which includes the laid back breastfeeding position with a lactation simulation model.
  Interventions: Behavioral: Breastfeeding position education with lactation simulation model
- Experimental: Upright breastfeeding position education group (Experimental): Breastfeeding education will be given to pregnant women in the upright breastfeeding position group, which includes the upright breastfeeding position with a lactation simulation model.
  Interventions: Behavioral: Breastfeeding position education with lactation simulation model
- No Intervention: Control Group (No Intervention): Mothers in the control group will receive routine hospital care

INTERVENTIONS:
Behavioral: Breastfeeding position education with lactation simulation model — pregnant women will receive training with a lactation simulation model once in the last trimester.The pregnant woman will wear the lactation simulation model during the education period and show what she has learned practically on the model.Mothers who have given birth will be supported to practice the breastfeeding position in the postpartum service.
  Arms: Experimental: Laid back breastfeding position education group; Experimental: Upright breastfeeding position education group

SUMMARY:
Planned for the purpose to evaluate, breast problems (nipple fissure, nipple pain), breastfeeding self-efficacy, breastfeeding success, and infant feeding attitude of mothers by given breastfeeding education with a laid back (semi-sitting or semi-lying) and upright position (sitting upright) using lactation simulation model.

DETAILED DESCRIPTION:
This study aims to increase breastfeeding success, breastfeeding self-efficacy and effective infant feeding, reduce breast problems, and to affect positively the mother's infant feeding attitude of breastfeeding positions taught to mothers in the antenatal period with the lactation simulation model. Also, it carried out to reveal the importance of midwife/nurse support and education that starts in the antenatal period and continues in the postpartum period, by increasing the adaptation of the mother to the breastfeeding process with the education given in the antenatal period, aims to contribute to the initiation and maintenance of breastfeeding. his study will be conducted as a randomized controlled experimental study. The population of the study will be primiparous pregnant women who applied to Kastamonu Education and Research Hospital between 01/05/2022-01/05/2023. The sample will consist of 105 pregnant women (35 pregnant women for each group) who met the inclusion criteria and accepted to participate in the study. The mothers in the experimental group will be trained with the lactation simulation model during the antenatal care follow-ups in the last trimester of their pregnancy (one group laid back and another group breastfeeding position education) and the necessary forms will be filled in their first interview, A second interview will be held within the first 24 hours after the birth, and the breastfeeding position taught to the mothers will be shown in practice by supporting the mother, and the necessary forms will be filled. The third meeting will be held between 7.-10. days of postpartum and the necessary forms will be filled. The mothers in the control group will be interviewed during the antenatal care follow-ups in the last trimester of their pregnancy. Mothers in the control group will receive routine care and routine breastfeeding education both in the prenatal and postnatal period. Necessary forms will be filled with the mothers in the control group by meeting in the first 24 hours and on the days 7th-10th. of postpartum. Personal information form, breastfeeding self-efficacy scale, Iowa infant feeding attitude scale, LATCH, visual comparison scale, postpartum breastfeeding follow-up form, breast problems evaluation form and IMDAT form will be used as data collection tools. Breastfeeding has numerous benefits for mother and baby. While it prevents many diseases such as otitis media, respiratory tract infections, obesity, sudden infant death syndrome, allergies and diabetes in infants, it neurodevelopmentally contributes positive effects to the development of the baby. Postpartum depression, cardiovascular diseases, diabetes, breast cancer, ovarian cancer and osteoporosis rates are lower in mothers who breastfeed for more than 1 year. The fact that there is less feeding cost contributes to the family economically.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women
* Primiparous
* Women aged 18-35 years
* Sign the informed consent form
* Those planning a vaginal birth
* Absence of a health problem that prevents breastfeeding
* Having a healthy baby at term

Exclusion Criteria:

* Diseases in which breastfeeding is a problem
* Baby with anomalies
* Cesarean births
* Patients admitted to neonatal intensive care

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women who are pregnancy
Enrollment: 105 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Iowa Infant Feeding Attitude Scale | Measurement for each group at the third encounter (10th day after birth).
  It is a scale that evaluates the attitudes of women towards breastfeeding and the choice of infant feeding method, as well as the duration of breastfeeding.The scale consists of a 5-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree) and 17 items. While 9 items in the scale affirm the issue of breastfeeding, 8 items contain positive statements about formula feeding. Formula nutrition items are scored in reverse (1=5, 2=4, 4=2 and 5=1). The total attitude score ranges from 17 (reflecting a positive attitude towards bottle feeding) to 85 points (reflecting a positive attitude towards breastfeeding). The scale has no cut-off value, high scores indicate a positive breastfeeding attitude. In the literature, those with a score between 70-85 were considered determined to breastfeed. If the score is between 49-69, the undecided group; Those with a score between 17-48 were accepted as having a tendency to feed with formula.
Breastfeeding Self-Efficacy Scale | Measurement for each group at the third encounter (10th day after birth).
  Breastfeeding self-efficacy levels of mothers and their self-confidence in breastfeeding are measured using the breastfeeding self-efficacy scale. The Breastfeeding Self-Efficacy Scale (short form) consists of 14 items that measure the mother's breastfeeding self-efficacy. The maximum score that can be obtained from the scale is 70, and the minimum score is 14.High scores from the scale indicate high breastfeeding self-efficacy. The scale is 5-point Likert type; 1 = Not at all sure, 2 = Not very sure, 3 = Sometimes I am sure, 4 = I am sure, 5 = I am very sure.
LATCH | Measurement for each group at the third encounter (10th day after birth).
  Observation and evaluation of mothers' breastfeeding success is measured using the LATCH scale.The LATCH Breastfeeding Diagnostic and Evaluation Scale is a scale filled by the researcher through observation.
  L: (Latch on the brest)) A: (Audible Swallowing) T: (Type of Nipple) C: (Comfort of Breast/ Nipple) H: (Hold/ Position)
  LATCH consists of the combination of the first letters of the English equivalent of the five criteria defined above. Each item is evaluated between 0-2 points. The lowest score that can be obtained from the entire scale is 0 and the highest score is 10. The scale has no breakpoints. The low score on the scale indicates the need for active intervention, support and follow-up after discharge in breastfeeding. The higher the LATCH Breastfeeding Diagnosis and Evaluation Scale score, the higher the success of breastfeeding.
Visual Analogue Scale | Measurement for each group at the third encounter (10th day after birth).
  It measures the severity of pain in individuals.This distance, which is usually measured in centimeters, is reported as "points". Numbers from 0 to 10 are written on the two ends of a 10 cm line on the parameter to be evaluated, and the patient is asked at what level of pain he is.The patient marks her own pain on a 10 cm ruler, with painlessness on one end and the most severe pain on the other. As the VAS value approaches 10, the pain is considered to be very severe, and as it approaches 0, the pain decreases.
IMDAT | Measurement for each group at the third encounter (10th day after birth).
  The amount of breast milk the baby receives is measured using the IMDAT scale.The form consists of 5 sections: the weight of the babies, their satisfaction, the frequency and characteristics of urinating and defecation, and the condition of the mother's breasts. With the form, the features of each situation are evaluated as 0, 1, 2 points, and the maximum total score that can be obtained is 10. A score of 8-10 is considered the best breast milk intake, and a score of 0-7 is considered insufficient.
Breast Problems Evaluation Form | Measurement for each group at the third encounter (10th day after birth).
  Problems such as pain, cracks and redness in the breast are measured using the breast evaluation form.The form consists of 9 questions questioning the breast problems of the mothers in the first 10 days postpartum. The form will be collected by the researcher through a face-to-face interview
Postpartum Breastfeeding Follow-Up Form | Measurement for each group at the third encounter (10th day after birth).
  This form was developed by the researcher by scanning the literature. The form consists of 13 questions questioning the postpartum breastfeeding status of mothers. The form will be collected by the researcher through a face-to-face interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Univercity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The research article will be shared after publication

REFERENCES:
- [Background] Coca KP, Marcacine KO, Gamba MA, Correa L, Aranha AC, Abrao AC. Efficacy of Low-Level Laser Therapy in Relieving Nipple Pain in Breastfeeding Women: A Triple-Blind, Randomized, Controlled Trial. Pain Manag Nurs. 2016 Aug;17(4):281-9. doi: 10.1016/j.pmn.2016.05.003. Epub 2016 Jun 27. PMID 27363734
- [Background] Colson S. Biological Nurturing: the laid-back breastfeeding revolution. Midwifery Today Int Midwife. 2012 Spring;(101):9-11, 66. No abstract available. PMID 22486009
- [Background] Mirghafourvand M, Kamalifard M, Ranjbar F, Gordani N. Relationship of breastfeeding self-efficacy with quality of life in Iranian breastfeeding mothers. J Matern Fetal Neonatal Med. 2018 Oct;31(20):2721-2728. doi: 10.1080/14767058.2017.1354368. Epub 2017 Jul 20. PMID 28728490
- [Background] Kestler-Peleg M, Shamir-Dardikman M, Hermoni D, Ginzburg K. Breastfeeding motivation and Self-Determination Theory. Soc Sci Med. 2015 Nov;144:19-27. doi: 10.1016/j.socscimed.2015.09.006. Epub 2015 Sep 8. PMID 26372935
- [Background] Kilci H, Coban A. The Correlation Between Breastfeeding Success in the Early Postpartum Period and the Perception of Self-Efficacy in Breastfeeding and Breast Problems in the Late Postpartum. Breastfeed Med. 2016 May;11:188-95. doi: 10.1089/bfm.2015.0046. Epub 2016 Mar 30. PMID 27027656
- [Background] McFadden A, Gavine A, Renfrew MJ, Wade A, Buchanan P, Taylor JL, Veitch E, Rennie AM, Crowther SA, Neiman S, MacGillivray S. Support for healthy breastfeeding mothers with healthy term babies. Cochrane Database Syst Rev. 2017 Feb 28;2(2):CD001141. doi: 10.1002/14651858.CD001141.pub5. PMID 28244064
- [Background] Milinco M, Travan L, Cattaneo A, Knowles A, Sola MV, Causin E, Cortivo C, Degrassi M, Di Tommaso F, Verardi G, Dipietro L, Piazza M, Scolz S, Rossetto M, Ronfani L; Trieste BN (Biological Nurturing) Investigators. Effectiveness of biological nurturing on early breastfeeding problems: a randomized controlled trial. Int Breastfeed J. 2020 Apr 5;15(1):21. doi: 10.1186/s13006-020-00261-4. PMID 32248838